CLINICAL TRIAL: NCT02137837
Title: Fulvestrant Alone Versus Fulvestrant and Everolimus Versus Fulvestrant, Everolimus and Anastrozole: A Phase III Randomized Placebo-Controlled Trial in Postmenopausal Patients
Brief Title: S1222 Trial (Everolimus, Anastrozole and Fulvestrant) in Post-Menopausal Stage IV Breast Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: AstraZeneca (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S1222
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Results first posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
Keywords: Metastatic breast cancer; Invasive breast carcinoma; estrogen receptor-positive breast cancer; HER2-negative breast cancer; Stage IV breast cancer; progesterone receptor-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Anastrozole; Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: fulvestrant + everolimus placebo + anastrozole placebo (Placebo Comparator): Patients receive an injection of fulvestrant in each buttock on Days 1 &15 for Cycle 1 and then Day 1 only for subsequent cycles. Patients also receive an oral placebo daily for both everolimus and anastrozole. This treatment regimen will continue until disease progression or toxicity.
  Interventions: Drug: Fulvestrant; Drug: Placebo - Anastrozole; Drug: Placebo - Everolimus
- Arm 2: fulvestrant + everolimus + anastrozole placebo (Experimental): Patients receive an injection of fulvestrant in each buttock on Days 1 &15 for Cycle 1 and then Day 1 only for subsequent cycles. Patients also receive an oral everolimus and an oral placebo for anastrozole daily. This treatment regimen will continue until disease progression or toxicity.
  Interventions: Drug: Fulvestrant; Drug: Everolimus; Drug: Placebo - Anastrozole
- Arm 3: fulvestrant + everolimus + anastrozole (Experimental): Patients receive an injection of fulvestrant in each buttock on Days 1 &15 for Cycle 1 and then Day 1 only for subsequent cycles. Patients also receive everolimus and anastrozole by mouth daily. This treatment regimen will continue until disease progression or toxicity.
  Interventions: Drug: Fulvestrant; Drug: Anastrozole; Drug: Everolimus

INTERVENTIONS:
Drug: Fulvestrant
  Other Names: Faslodex; NSC-719276
Drug: Anastrozole
  Other Names: Arimidex; NSC-719344
  Arms: Arm 3: fulvestrant + everolimus + anastrozole
Drug: Everolimus
  Other Names: Afinitor; Zortress; NSC-733504
  Arms: Arm 2: fulvestrant + everolimus + anastrozole placebo; Arm 3: fulvestrant + everolimus + anastrozole
Drug: Placebo - Anastrozole
  Arms: Arm 1: fulvestrant + everolimus placebo + anastrozole placebo; Arm 2: fulvestrant + everolimus + anastrozole placebo
Drug: Placebo - Everolimus
  Arms: Arm 1: fulvestrant + everolimus placebo + anastrozole placebo

SUMMARY:
This randomized Phase III trial studies how well the combination of fulvestrant and everolimus together or the combination of anastrozole, fulvestrant and everolimus together, improve progression-free survival (PFS) versus fulvestrant alone.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To test the benefit of interfering with the function of the estrogen receptor (ER) and providing downstream target inhibition (PI3K/AKT/mTOR) with a combination of optimal dose fulvestrant and everolimus (Arm 2) to improve progression-free survival compared to the optimal dose fulvestrant alone (Arm 1).
* To test the benefit of adding the non-steroidal aromatase inhibitor anastrozole to optimal dose fulvestrant and everolimus (Arm 3) in order to improve progression free survival over optimal dose fulvestrant (Arm 1).

Secondary

* To compare progression-free survival among those receiving fulvestrant + everolimus + anastrozole (Arm 3) versus fulvestrant + everolimus (Arm 2).
* To compare overall survival among the treatment arms in post-menopausal patients with hormone-receptor positive (HR+) Stage IV breast cancer.
* To assess and compare toxicities, feasibility and compliance among the study regimens.
* To compare response rates and clinical benefit rates among the study regimens.
* To test molecular determinants of response to endocrine therapy and everolimus in circulating tumor cells:

  1. CTC-Endocrine Therapy Index (CTC ETI) on the CellSearch® platform.
  2. CTC-Next Generation Sequencing Analysis (CTC-NGS) of single cells captured on the HD-CTC® platform.

OUTLINE:

This is a multicenter study. Patients will be stratified according to the following factors:

* Measurable versus evaluable non-measurable disease
* Prior adjuvant hormonal therapy completed more than 5 years ago vs. prior adjuvant hormonal therapy completed 1-5 years ago vs. de novo presentation of metastatic disease or no prior adjuvant hormonal therapy.

ARMS:

* Arm 1: fulvestrant + placebo (everolimus) + placebo (anastrozole)
* Arm 2: fulvestrant + everolimus + placebo (anastrozole)
* Arm 3: fulvestrant + everolimus + anastrozole

Blood and tissue samples are collected for correlative science studies.

After completion of study treatment, patients are followed up every 6 months for 2 years and then yearly thereafter for 5 years.

ELIGIBILITY:
* Patients must have a histologically confirmed diagnosis of invasive breast carcinoma with positive estrogen and/or progesterone receptor status, and negative human epidermal growth factor receptor (HER-2), for whom endocrine therapy is planned.
* The HER-2 test result is negative (and should be reported as such), if a single test (or all tests)performed in a tumor specimen show:

  * Immunohistochemistries (IHC) 1+ negative or IHC 0 negative or
  * in situ hybridization (ISH) negative using a single probe ISH or dual probe ISH.
* Estrogen receptor (ER) and progesterone receptor (PgR) positivity must be assessed according to American Society of Clinial Oncology (ASCO)/College of American Physicians (CAP) guidelines as either ER or PR ≥ 1% positive nuclear staining. If HER2 IHC is 2+, an evaluation for gene amplification must be performed and the gene must not be amplified. Gene amplification evaluation is not required if evaluation by IHC is 0 or 1+ by institutional standards.
* Patients must be post-menopausal women with a confirmed diagnosis of metastatic breast cancer (M1). Pathologic confirmation of histology is preferable. In the case of bone metastases only, biopsy-proven metastatic disease of solitary site, or multiple sites of involvement are required. Post-menopausal is defined by one of the following criteria as per National Comprehensive Cancer Network (NCCN) guidelines Version 3. 2013:

  * Prior bilateral oophorectomy and/or hysterectomy
  * Patients ≥ 60 years of age
  * Patients < 60 years of age and amenorrheic for ≥ 12 months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression and follicle-stimulating hormone (FSH) and estradiol in the post-menopausal range
  * Patients < 60 years of age taking tamoxifen or toremifene must have FSH and plasma estradiol levels within post-menopausal ranges
* Patients must have measurable or evaluable disease. Patients must have a chest and abdominal computerized tomography (CT) and bone scan within 28 days prior to registration. All scans needed for assessment of measurable disease must be performed within 28 days prior to registration. Evaluable disease must be assessed within 28 days prior to registration
* Patients with a history of prior chemotherapy or hormone therapy or immunotherapy for recurrent or metastatic disease are NOT eligible. Prior adjuvant or neoadjuvant chemotherapy if completed more than 12 months prior to registration is acceptable. Any number of prior hormonal therapy regimens for the adjuvant setting but not for metastatic or recurrent disease is allowed; prior adjuvant or neoadjuvant treatment with an aromatase inhibitor (e.g. anastrozole, letrozole, exemestane) is allowed, if completed more than 12 months prior to randomization.
* Patients who have taken luteinizing hormone-releasing hormone (LHRH) analogue as adjuvant therapy are eligible provided they have a) discontinued such therapy at least 12 months prior to registration AND b) have not resumed their menstrual periods.
* Patients must not have had prior exposure to fulvestrant or mTOR inhibitors (e.g., rapamycin, everolimus, temsirolimus, deforolimus). Concurrent bisphosphonate therapy is allowed. Patients must not have prior treatment with any investigational drug within 28 days prior to registration and must not be planning to receive any other investigational drug for the duration of the study.
* Patients must have an International Normalized Ratio (INR) ≤ 1.6 within 28 days prior to registration.
* Patients must have adequate bone marrow function, as defined by Absolute Neutrophil Count (ANC) of ≥ 1,500/mL, hemoglobin ≥ 9 g/dL and a peripheral platelet count ≥ 100,000/ mL, all within 28 days prior to registration.
* Patients must have adequate hepatic function obtained within 28 days prior to registration and documented by all of the following:

  * Bilirubin ≤ 1.5 mg/dL (or ≤ 3.0 mg/dL if due to Gilbert's Syndrome)
  * alanine aminotransferase (ALT) (SGPT) and aspartate aminotransferase (AST) (SGOT) ≤ 2.5 x Institutional Upper Limit of Normal (IULN), or ≤ 5 x IULN if hepatic metastases are present.
* Patients must have adequate renal function with serum creatinine level ≤ IULN within 28 days prior to registration.
* Patients must have a fasting cholesterol ≤ 300 mg/dL and triglycerides ≤ 2.5 x IULN obtained within 28 days prior to registration. Patients may be on lipid lowering agents to reach these values.
* Patients must have a complete history and physical examination within 28 days prior to registration.
* Patients with bleeding diathesis (i.e., disseminated intravascular coagulation [DIC], clotting factor deficiency) or long-term anti-coagulant therapy (other than antiplatelet therapy) are NOT eligible.
* Patients with presence of life-threatening metastatic visceral disease, defined as extensive hepatic involvement, or any degree of brain or leptomeningeal involvement (past or present), or symptomatic pulmonary lymphangitic spread are not eligible. Patients with discrete pulmonary parenchymal metastases are eligible, provided their respiratory function is not significantly compromised as a result of disease in the opinion of the investigator.
* Patients must have a performance status of 0 - 2 by Zubrod criteria.
* Patients must not have any Grade III/IV cardiac disease as defined by the New York Heart Association Criteria (i.e., patients with cardiac disease resulting in marked limitation of physical activity or resulting in inability to carry on any physical activity without discomfort), unstable angina pectoris, myocardial infarction within 6 months, or serious uncontrolled cardiac arrhythmia.
* Patients must not have uncontrolled diabetes (defined as an Hg A1C >7% within 28 days prior to registration).
* Patients must not have an organ allograft or other history of immune compromise. Patients must not be receiving chronic, systemic treatment with corticosteroids or other immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Patients known to be HIV positive may be enrolled if baseline CD4 count is > 500 cells/mm3 AND not taking anti-retroviral therapy. Patients with known chronic or active hepatitis are not eligible. Patients must not have any known uncontrolled underlying pulmonary disease.
* Patients must be able to take oral medications. Patient may not have any impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).
* Patients must not have received immunization with an attenuated live vaccine (e.g. intranasal influenza, MMR, oral polio, varicella, zoster, yellow fever and BCG vaccines) within seven days prior to registration nor have plans to receive such vaccination while on protocol treatment.
* Patients must not have taken within 14 days prior to registration, be taking, nor plan to take while on protocol treatment, strong CYP3A4 inhibitors, and/or CYP3A4 inducers.
* No other prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer or other cancer for which the patient has been disease-free for 5 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-05; Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Halle Moore, M.D., Study Chair — The Cleveland Clinic
Locations (223):
- United States (223):
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Virginia G. Piper Cancer Center, Scottsdale, Arizona
  - University of Arizona Cancer Center - Orange Grove, Tucson, Arizona
  - University of Arizona Cancer Center - North Campus, Tucson, Arizona
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - University of Arizona Medical Center - Univ Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Providence St. Joseph Medical Ctr/Disney Family CC, Burbank, California
  - City of Hope-Corona, Corona, California
  - City of Hope National Medical Center, Duarte, California
  - City of Hope Antelope Valley, Lancaster, California
  - Bay Area Tumor Institute, Oakland, California
  - Summit Medical Center, Oakland, California
  - Epic Care - Oakland, Oakland, California
  - City of Hope South Pasadena, South Pasadena, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - St. Francis Hospital and Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Sacred Heart Hospital, Pensacola, Florida
  - Cleveland Clinic - Weston, Weston, Florida
  - South Georgia Medical Center - Pearlman Cancer Ctr, Valdosta, Georgia
  - Oncare Hawaii Inc-POB I, Honolulu, Hawaii
  - Oncare Hawaii, Inc - POB II, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Oncare Hawaii, Inc - Kuakini, Honolulu, Hawaii
  - Oncare Hawaii, Inc - Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Oncare Hawaii, Inc - Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - St. Alphonsus Regional Medical Center, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Centralia Oncology Clinic, Centralia, Illinois
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Kishwaukee Community Hospital, DeKalb, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Loyola University Stritch School of Medicine, Maywood, Illinois
  - Marjorie Weinberg Cancer Center, Melrose Park, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas - Independence, Independence, Kansas
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas - Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates in Women's Health, Wichita, Kansas
  - Cancer Center of Kansas - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - De Soto Regional Medical Center, Mansfield, Louisiana
  - University Health Conway, Monroe, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Winchester Hospital, Winchester, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Oakwood Healthcare, Inc., Dearborn, Michigan
  - Wayne State University Medical Center, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - William Beaumont Hospital-Grosse Pointe, Grosse Pointe, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Health System, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - St Joseph Mercy Hospital - Oakland, Pontiac, Michigan
  - St. Joseph Mercy Port Huron, Port Huron, Michigan
  - Beaumont Children's Hospital-Royal Oak, Royal Oak, Michigan
  - Beaumont NCI Community Oncology Research Program, Royal Oak, Michigan
  - St. Mary's Health System, Saginaw, Michigan
  - Beaumont Hospital, Troy Campus, Troy, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Ctr-Carrie J. Babb Cancer Ctr, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - St. Francis Medical Center, Cape Girardeau, Missouri
  - Mercy Hospital - Joplin, Joplin, Missouri
  - Mercy Clinic Care and Hematology - Rolla, Rolla, Missouri
  - PCRMC Bond Clinic, Rolla, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - St. Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Christian Hospital, St Louis, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Community Hosp and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare West Campus, Great Falls, Montana
  - St. Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - St. Patrick Hospital, Missoula, Montana
  - CHI Health Good Samaritan Hospital, Kearney, Nebraska
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R. Pardee Memorial Hospital, Hendersonville, North Carolina
  - Park Ridge Health, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Cleveland Clinic Cancer Center - Beachwood, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - VA Medical Center - Cincinnati, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center - Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - The Mark H. Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Good Samaritan Hospital and Health Center, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - VA Medical Center - Dayton, Dayton, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center - Independence, Independence, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Cleveland Clinic Cancer Center - Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Inc., Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Cleveland Clinic Strongsville Family Health Center, Strongsville, Ohio
  - Upper Valley Medical Centers, Troy, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - St. Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic Cancer Center - Wooster, Wooster, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - St. Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - McLeod Regional Medical Center, Florence, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Cancer, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology, Bristol, Tennessee
  - Wellmont Medical Assoc Onc and Hem-Johnson City, Johnson City, Tennessee
  - Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Wellmont Medical Assoc Onc and Hem-Kingsport, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - University of Utah Medical Center, Salt Lake City, Utah
  - Southwest Virginia Cancer Center, Norton, Virginia
  - Island Hospital, Anacortes, Washington
  - Auburn Regional Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Swedish Cancer Inst-Eastside Oncology Hematoly, Bellevue, Washington
  - PeaceHealth St. Joseph Medical Center, Bellingham, Washington
  - Swedish Medical Center - Edmonds, Edmonds, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Ctrs-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - PeaceHealth St. John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Ctrs-Puyallup, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Pacific Cancer Research Consortium NCORP, Seattle, Washington
  - Pacific Medical Center - First Hill, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Swedish Medical Center - Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Tacoma/Valley Radiation Oncology Ctrs-Jackson Hill, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Ctrs-Saint Joe's, Tacoma, Washington
  - Multicare Health System, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center - Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Fulvestrant + Everolimus Placebo + Anastrozole Placebo: Participants receive an injection of fulvestrant in each buttock on Days 1 &15 for Cycle 1 and then Day 1 only for subsequent cycles. Participants also receive an oral placebo daily for both everolimus and anastrozole. This treatment regimen will continue until disease progression or toxicity.
  Fulvestrant
  Placebo - Anastrozole
  Placebo - Everolimus
- Arm 2: Fulvestrant + Everolimus + Anastrozole Placebo: Participants receive an injection of fulvestrant in each buttock on Days 1 &15 for Cycle 1 and then Day 1 only for subsequent cycles. Participants also receive an oral everolimus and an oral placebo for anastrozole daily. This treatment regimen will continue until disease progression or toxicity.
  Fulvestrant
  Everolimus
  Placebo - Anastrozole
- Arm 3: Fulvestrant + Everolimus + Anastrozole: Participants receive an injection of fulvestrant in each buttock on Days 1 &15 for Cycle 1 and then Day 1 only for subsequent cycles. Participants also receive everolimus and anastrozole by mouth daily. This treatment regimen will continue until disease progression or toxicity.
  Fulvestrant
  Anastrozole
  Everolimus
Period: Overall Study
Arm/Group | Arm 1: Fulvestrant + Everolimus Placebo + Anastrozole Placebo | Arm 2: Fulvestrant + Everolimus + Anastrozole Placebo | Arm 3: Fulvestrant + Everolimus + Anastrozole
Started | 13 | 12 | 12
Received Protocol Therapy | 13 | 11 | 12
Completed | 0 | 0 | 0
Not Completed | 13 | 12 | 12
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Refusal unrelated to adverse event | 2 | 2 | 1
Not completed — Progression/relapse | 9 | 7 | 7
Not completed — Not protocol specified | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Eligible participants randomized to study arms
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Fulvestrant + Everolimus Placebo + Anastrozole Placebo | Arm 2: Fulvestrant + Everolimus + Anastrozole Placebo | Arm 3: Fulvestrant + Everolimus + Anastrozole | Total
Number analyzed (Participants) | 13 | 12 | 12 | 37
Age, Continuous [Median (Full Range); unit: years] | 63.4 [54.9 to 74.0] | 62.6 [45.6 to 87.9] | 60.5 [48.2 to 69.5] | 62.0 [45.6 to 87.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 12 | 37
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 12 | 10 | 12 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 3 | 5
  White | 9 | 10 | 9 | 28
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 0 | 2
Disease [Number; unit: participants]
  Measurable | 9 | 10 | 9 | 28
  Evaluable non-measurable disease | 4 | 2 | 3 | 9
Prior Hormone [Count of Participants; unit: Participants]
  Prior adjuvant hormonal therapy completed >5 years ago | 3 | 1 | 2 | 6
  Prior adjuvant hormonal therapy completed 1-5 years ago | 4 | 5 | 6 | 15
  De novo presentation of metastatic disease or no prior adjuvant hormonal therapy | 6 | 6 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (Fulvestrant vs Fulvestrant + Everolimus )
Description: From date of registration to date of first documentation of progression or death due to any cause. Participants last known to be alive are censored at date of last contact.
Time Frame: up to 5 years
Population: Eligible participants randomized to study arms. This includes 1 participant on arm 2 who did not receive protocol treatment and is assumed to be a non-responder for response assessment.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm 1: Fulvestrant + Everolimus Placebo + Anastrozole Placebo: Participants receive an injection of fulvestrant in each buttock on Days 1 &15 for Cycle 1 and then Day 1 only for subsequent cycles. Participants also receive an oral placebo daily for both everolimus and anastrozole. This treatment regimen will continue until disease progression or toxicity. (Note: after study unblinding at time of permanent study closure, participants on this arm received fulvestrant without continuing placebos.)
  Fulvestrant
  Placebo - Anastrozole
  Placebo - Everolimus
- Arm 2: Fulvestrant + Everolimus + Anastrozole Placebo: Participants receive an injection of fulvestrant in each buttock on Days 1 &15 for Cycle 1 and then Day 1 only for subsequent cycles. Participants also receive an oral everolimus and an oral placebo for anastrozole daily. This treatment regimen will continue until disease progression or toxicity. (Note: after study unblinding at time of permanent study closure, participants on this arm received fulvestrant and unblinded everolimus without continuing placebos.)
  Fulvestrant
  Everolimus
  Placebo - Anastrozole
Arm/Group | Arm 1: Fulvestrant + Everolimus Placebo + Anastrozole Placebo | Arm 2: Fulvestrant + Everolimus + Anastrozole Placebo
Number analyzed (Participants) | 13 | 12
months | 14.0 [NA to NA] — Confidence intervals not calculated due to small sample size | 11.3 [NA to NA] — Confidence intervals not calculated due to small sample size

2. Primary Outcome: Progression-free Survival (Fulvestrant Versus Fulvestrant + Everolimus + Anastrozole)
Description: From date of registration to date of first documentation of progression or death due to any cause. Participants last known to be alive without report of progression are censored at date of last contact.
Time Frame: up to 5 years
Population: Eligible participants who were randomized to study arms and received protocol therapy
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm 3: Fulvestrant + Everolimus + Anastrozole: Participants receive an injection of fulvestrant in each buttock on Days 1 &15 for Cycle 1 and then Day 1 only for subsequent cycles. Participants also receive everolimus and anastrozole by mouth daily. This treatment regimen will continue until disease progression or toxicity. (Note: after study unblinding at time of permanent study closure, participants on this arm received fulvestrant and unblinded everolimus and anastrozole.)
  Fulvestrant
  Anastrozole
  Everolimus
Arm/Group | Arm 1: Fulvestrant + Everolimus Placebo + Anastrozole Placebo | Arm 3: Fulvestrant + Everolimus + Anastrozole
Number analyzed (Participants) | 13 | 12
months | 14.0 [NA to NA] — Confidence intervals not calculated due to small sample size | 9.9 [NA to NA] — Confidence intervals not calculated due to small sample size

3. Secondary Outcome: Progression Free Survival (Fulvestrant + Everolimus vs Fulvestrant + Everolimus + Anastrozole)
Description: as for outcome 2
Time Frame: up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 2: Fulvestrant + Everolimus + Anastrozole Placebo | Arm 3: Fulvestrant + Everolimus + Anastrozole
Number analyzed (Participants) | 12 | 12
months | 11.3 [NA to NA] — Confidence intervals not calculated due to small sample size | 9.90 [NA to NA] — Confidence intervals not calculated due to small sample size

4. Secondary Outcome: Overall Survival
Description: From date of registration to date of death due to any cause. Participants last known to be alive without report of progression are censored at date of last contact.
Time Frame: up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: Fulvestrant + Everolimus Placebo + Anastrozole Placebo | Arm 2: Fulvestrant + Everolimus + Anastrozole Placebo | Arm 3: Fulvestrant + Everolimus + Anastrozole
Number analyzed (Participants) | 13 | 12 | 12
months | 46.8 [NA to NA] — Confidence intervals not calculated due to small sample size | 56.6 [NA to NA] — Confidence intervals not calculated due to small sample size | 33.6 [NA to NA] — Confidence intervals not calculated due to small sample size

5. Secondary Outcome: Number of Patients With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE Version 4.0. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Duration of treatment and follow up until death or 5 years post registration
Population: Eligible participants who received at least one dose of protocol treatment.
Measure: Number; unit: Participants
Groups:
- Arm 1: Fulvestrant + Everolimus Placebo + Anastrozole Placebo: Participants receive an injection of fulvestrant in each buttock on Days 1 & 15 for Cycle 1 and then Day 1 only for subsequent cycles. Participants also receive an oral placebo daily for both everolimus and anastrozole. This treatment regimen will continue until disease progression or toxicity. (Note: after study unblinding at time of permanent study closure, participants on this arm received fulvestrant without continuing placebos.)
  Fulvestrant
  Placebo - Anastrozole
  Placebo - Everolimus
- Arm 2: Fulvestrant + Everolimus + Anastrozole Placebo: Participants receive an injection of fulvestrant in each buttock on Days 1 & 15 for Cycle 1 and then Day 1 only for subsequent cycles. Participants also receive an oral everolimus and an oral placebo for anastrozole daily. This treatment regimen will continue until disease progression or toxicity. (Note: after study unblinding at time of permanent study closure, participants on this arm received fulvestrant and unblinded everolimus without continuing placebos.)
  Fulvestrant
  Everolimus
  Placebo - Anastrozole
- Arm 3: Fulvestrant + Everolimus + Anastrozole: Participants receive an injection of fulvestrant in each buttock on Days 1 & 15 for Cycle 1 and then Day 1 only for subsequent cycles. Participants also receive everolimus and anastrozole by mouth daily. This treatment regimen will continue until disease progression or toxicity. (Note: after study unblinding at time of permanent study closure, participants on this arm received fulvestrant and unblinded everolimus and anastrozole.)
  Fulvestrant
  Anastrozole
  Everolimus
Arm/Group | Arm 1: Fulvestrant + Everolimus Placebo + Anastrozole Placebo | Arm 2: Fulvestrant + Everolimus + Anastrozole Placebo | Arm 3: Fulvestrant + Everolimus + Anastrozole
Number analyzed (Participants) | 13 | 11 | 12
Participants
  Abdominal pain | 0 | 1 | 0
  Anorexia | 0 | 1 | 1
  Aspartate aminotransferase increased | 0 | 1 | 0
  Dehydration | 0 | 2 | 1
  Diarrhea | 0 | 1 | 0
  Fatigue | 0 | 2 | 0
  Flu like symptoms | 0 | 1 | 0
  Generalized muscle weakness | 0 | 1 | 0
  Hyperglycemia | 0 | 1 | 0
  Hypertension | 0 | 2 | 2
  Hypocalcemia | 0 | 1 | 0
  Hypokalemia | 0 | 2 | 1
  Hyponatremia | 0 | 1 | 0
  Hypophosphatemia | 0 | 1 | 0
  Hypotension | 0 | 0 | 1
  Localized edema | 0 | 1 | 0
  Lymphocyte count decreased | 0 | 1 | 0
  Mucositis oral | 0 | 0 | 1
  Neutrophil count decreased | 0 | 2 | 0
  Rash maculo-papular | 0 | 0 | 1
  Resp, thoracic and mediastinal disorders - Other | 0 | 1 | 0
  Sore throat | 0 | 0 | 1
  Thromboembolic event | 0 | 0 | 1
  Vomiting | 0 | 1 | 0
  White blood cell decreased | 0 | 1 | 0

6. Secondary Outcome: Response Rate
Description: Proportion of participants who have confirmed or unconfirmed partial or complete response to therapy
Time Frame: assessed every 12 weeks, up to 5 years
Population: Eligible participants with measurable disease.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Fulvestrant + Everolimus Placebo + Anastrozole Placebo | Arm 2: Fulvestrant + Everolimus + Anastrozole Placebo | Arm 3: Fulvestrant + Everolimus + Anastrozole
Number analyzed (Participants) | 9 | 10 | 9
percentage of participants | 22 | 60 | 44

7. Secondary Outcome: Clinical Benefit Rate
Description: Proportion of participants who have confirmed and unconfirmed partial response, complete response or stable disease.
Time Frame: assessed every 12 weeks, up to 5 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Fulvestrant + Everolimus Placebo + Anastrozole Placebo | Arm 2: Fulvestrant + Everolimus + Anastrozole Placebo | Arm 3: Fulvestrant + Everolimus + Anastrozole
Number analyzed (Participants) | 13 | 12 | 12
percentage of participants | 69 | 83 | 67

8. Secondary Outcome: Molecular Determinants of Response in Circulating Tumor Cells: CTC-ETI
Description: CTC-Endocrine Therapy Index (CTC-ETI) on the CellSearch® platform. Based on enumeration of CTC/7.5 mL of whole blood, with >= 5 being elevated. (Due to limited samples collected, full analysis was not able to be performed as planned, so outcome measure reported here is number with elevated Day 1 CTC.)
Time Frame: Day 1, Day 29, time of progression (Day 29 to be collected only if Day 1 CTC was elevated.)
Population: Participants with Day 1 whole blood specimen submitted.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Fulvestrant + Everolimus Placebo + Anastrozole Placebo | Arm 2: Fulvestrant + Everolimus + Anastrozole Placebo | Arm 3: Fulvestrant + Everolimus + Anastrozole
Number analyzed (Participants) | 5 | 5 | 3
Participants | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 5 years post registration
Description: 36 participants who were eligible and received protocol therapy were assessed for AEs.
Groups:
- Arm 1: Fulvestrant + Everolimus Placebo + Anastrozole Placebo: Participants receive an injection of fulvestrant in each buttock on Days 1 & 15 for Cycle 1 and then Day 1 only for subsequent cycles. Participants also receive an oral placebo daily for both everolimus and anastrozole. This treatment regimen will continue until disease progression or toxicity.
  Fulvestrant
  Placebo - Anastrozole
  Placebo - Everolimus
- Arm 2: Fulvestrant + Everolimus + Anastrozole Placebo: Participants receive an injection of fulvestrant in each buttock on Days 1 & 15 for Cycle 1 and then Day 1 only for subsequent cycles. Participants also receive an oral everolimus and an oral placebo for anastrozole daily. This treatment regimen will continue until disease progression or toxicity.
  Fulvestrant
  Everolimus
  Placebo - Anastrozole
- Arm 3: Fulvestrant + Everolimus + Anastrozole: Participants receive an injection of fulvestrant in each buttock on Days 1 & 15 for Cycle 1 and then Day 1 only for subsequent cycles. Participants also receive everolimus and anastrozole by mouth daily. This treatment regimen will continue until disease progression or toxicity.
  Fulvestrant
  Anastrozole
  Everolimus
Arm/Group | Arm 1: Fulvestrant + Everolimus Placebo + Anastrozole Placebo | Arm 2: Fulvestrant + Everolimus + Anastrozole Placebo | Arm 3: Fulvestrant + Everolimus + Anastrozole
All-Cause Mortality (participants affected / at risk) | 8/13 | 6/12 | 6/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 13/13 | 11/11 | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Fulvestrant + Everolimus Placebo + Anastrozole Placebo (N=13) | Arm 2: Fulvestrant + Everolimus + Anastrozole Placebo (N=11) | Arm 3: Fulvestrant + Everolimus + Anastrozole (N=12)
Anemia (Blood and lymphatic system disorders) | 4 | 8 | 6
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1
Cardiac disorders-Other (Cardiac disorders) | 0 | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 3 | 0
Ear and labyrinth disorders-Other (Ear and labyrinth disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
External ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Blurred vision (Eye disorders) | 0 | 1 | 1
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Eye disorders-Other (Eye disorders) | 2 | 1 | 0
Floaters (Eye disorders) | 0 | 1 | 0
Watering eyes (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 1
Anal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 6 | 7
Dental caries (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 5 | 4
Dry mouth (Gastrointestinal disorders) | 3 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 2 | 0
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 1 | 2 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 7 | 8
Nausea (Gastrointestinal disorders) | 5 | 6 | 4
Oral pain (Gastrointestinal disorders) | 2 | 2 | 3
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 4
Chills (General disorders) | 1 | 2 | 1
Edema face (General disorders) | 0 | 1 | 0
Edema limbs (General disorders) | 4 | 6 | 3
Fatigue (General disorders) | 10 | 10 | 7
Fever (General disorders) | 3 | 3 | 1
Flu like symptoms (General disorders) | 0 | 1 | 1
General disorders and admin site conditions - Other (General disorders) | 1 | 3 | 0
Injection site reaction (General disorders) | 2 | 1 | 0
Localized edema (General disorders) | 0 | 3 | 1
Malaise (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 2 | 1
Pain (General disorders) | 4 | 2 | 3
Allergic reaction (Immune system disorders) | 1 | 1 | 0
Immune system disorders-Other (Immune system disorders) | 0 | 2 | 0
Infections and infestations-Other (Infections and infestations) | 1 | 4 | 2
Mucosal infection (Infections and infestations) | 0 | 0 | 1
Rhinitis infective (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 1
Upper respiratory infection (Infections and infestations) | 2 | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 6 | 3
Alkaline phosphatase increased (Investigations) | 3 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 7 | 4
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Cholesterol high (Investigations) | 4 | 10 | 5
Creatinine increased (Investigations) | 0 | 1 | 2
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1 | 0
INR increased (Investigations) | 1 | 0 | 0
Investigations-Other (Investigations) | 0 | 2 | 1
Lipase increased (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 7 | 4
Neutrophil count decreased (Investigations) | 0 | 3 | 1
Platelet count decreased (Investigations) | 1 | 4 | 4
Weight gain (Investigations) | 1 | 1 | 2
Weight loss (Investigations) | 2 | 6 | 3
White blood cell decreased (Investigations) | 0 | 7 | 4
Anorexia (Metabolism and nutrition disorders) | 3 | 7 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 1
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 8 | 7 | 5
Hypernatremia (Metabolism and nutrition disorders) | 0 | 2 | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4 | 8 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 7 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 2 | 5 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 4 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 5 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 1
Dysesthesia (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 6 | 0
Headache (Nervous system disorders) | 4 | 4 | 5
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Nervous system disorders-Other (Nervous system disorders) | 0 | 2 | 0
Paresthesia (Nervous system disorders) | 0 | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 2 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 5 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2 | 1
Depression (Psychiatric disorders) | 2 | 0 | 1
Insomnia (Psychiatric disorders) | 3 | 3 | 2
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 1 | 0
Renal and urinary disorders-Other (Renal and urinary disorders) | 1 | 1 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 1 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 1 | 2
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 0 | 2 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal pain (Reproductive system and breast disorders) | 1 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 3 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 4 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 4 | 3
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0
Hot flashes (Vascular disorders) | 6 | 6 | 5
Hypertension (Vascular disorders) | 2 | 5 | 4
Hypotension (Vascular disorders) | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 1
Vascular disorders-Other (Vascular disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/37/NCT02137837/Prot_SAP_ICF_000.pdf